CLINICAL TRIAL: NCT07032181
Title: The Effect of Virtual Reality and Guided Imagery Method Used During Blood Sampling on Pain, Fear
Brief Title: The Effect of Non-pharmacological Methods on Pain, Fear
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Negarin Akbari, Assisstant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025.167.IRB2.075
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Children; Pain; Fear; Pediatric ALL
Keywords: Pediatric; Pain; Fear; Children; Blood Sampling
MeSH Terms: conditions — Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Imagery (Experimental): To implement the guided imagery method, a text titled "A Walk in the Forest" will be used. The text includes descriptions of living and non-living elements in the forest to help the child imagine taking a walk in a forest. It is designed to engage the child's physical senses through sensory language, encouraging a vivid mental experience.One minute before the blood collection procedure, the child will be given headphones and the audio recording will be started.
  The prepared text was recorded in a studio with the support of a professional audio recording specialist. The narration was performed by a professional voice actor specializing in voice work, who read the text in a calm and gentle tone. In the background, soft and slow-paced music was played, and nature sound effects-such as bird chirping, rustling leaves, and flowing water-were added at various points to match the flow of the text. The total duration of the audio recording is 2 minutes and 35 seconds.
  Interventions: Procedure: Virtual reality, guided imagery
- Virtual Reality (Experimental): Virtual reality (VR) glasses will be used in this study. A video or game compatible with a mobile phone will be loaded onto the device, placed in the front compartment of the VR glasses, and the cover will be closed. The glasses will then be positioned on the child's head. When selecting the VR glasses, attention will be given to choosing lightweight and child-friendly models.
  In the Virtual Reality Glasses group, unlike the Guided Imagery group, the child will wear VR glasses and watch a video titled "A Walk in the Forest", which was created using artificial intelligence.One minute before the blood collection procedure, the child will be start.
  Interventions: Procedure: Virtual reality, guided imagery
- Control (No Intervention): For the children in the control group, only a routine blood collection procedure will be performed, and they will receive only a standard explanation related to the procedure.

INTERVENTIONS:
Procedure: Virtual reality, guided imagery — Before the procedure, children will be informed via the Child Consent Form, and parents through the Informed Consent Form. Verbal and written consents will be obtained, and data will be recorded in the Child Patient Introductory Information Form. Pre-procedural pain will be assessed using the Faces Pain Scale-Revised scale, and the child will mark their pain. Parents will use the VAS scale for pain assessment. The CFS scale will be explained to both the child and parent to assess the child's fear. A pulse oximeter will measure SPO2 and pulse one minute before the procedure.
  The blood collection procedure will be performed by an experienced nurse, and heart rate and oxygen saturation will be recorded in the Application Record Form.
  After the procedure, measurements will be taken immediately after the procedure and one minute later.
  Children will mark their pain and fear levels on the FPS-R and CFS scales. Parents and observers will also assess the child's pain (VAS) and fear (CFS).
  Arms: Guided Imagery; Virtual Reality

SUMMARY:
This randomized controlled experimental study aims to evaluate the effectiveness of guided imagery and virtual reality (VR) in reducing pain and fear in children during blood draw procedures. The sample will consist of children aged 8-14 who meet the inclusion criteria and present to the Koç Hospital Pediatric Clinic Blood Drawing Room. After informing the children and their parents about the study, written and verbal consents will be obtained. Participants will then be randomly assigned into one of three groups-two experimental (guided imagery and VR) and one control-using a random number list generated via Excel.

Pre-procedure: Prior to the intervention, children and parents will be informed using consent forms. Demographic and baseline data will be collected using the Child Patient Introductory Information Form. Pain will be assessed with the Faces Pain Scale-Revised (FPS-R) by the child and the Visual Analog Scale (VAS) by the parent and observer. Fear will be evaluated using the Children's Fear Scale (CFS), self-rated by the child and assessed by the parent/observer. A pulse oximeter will be attached to measure baseline pulse and oxygen saturation (SpO2) levels starting 1 minute before the procedure.

Guided Imagery Group: Children will listen to an audio recording titled "A Walk in the Forest" using headphones. They will be instructed to close their eyes and imagine the scene described, focusing on the sound to facilitate distraction. The audio will start 1 minute prior to the procedure.

Virtual Reality Group: Children in this group will wear VR glasses and watch an immersive AI-generated video of "A Walk in the Forest." This aims to provide a more interactive distraction during the blood draw.

Control Group: Children will undergo routine blood draw procedures with no additional distraction techniques. The procedure will be explained as usual.

Procedure: A trained nurse will perform all blood draws. During the procedure, SpO2 and pulse data will be recorded. Post-procedure, these will also be documented immediately and 1 minute after the intervention.

Post-procedure: After the procedure, FPS-R and CFS will be used again by children to assess pain and fear. Parents and observers will complete VAS and CFS to evaluate observed pain and fear. Headphones or VR glasses will be removed following the final measurement.

DETAILED DESCRIPTION:
Randomization: Children aged 8 to 14, who meet the sample selection criteria and visit the blood collection room of the Koç Hospital Pediatric Clinic, will be introduced to the research. Information about the study will be provided, and written and verbal consent will be obtained from the children and their parents who volunteer to participate. Subsequently, the researcher will perform the randomization, assigning the children into three different groups: two experimental groups and one control group. A random number set generated using the Excel program will be used for randomization.

Pre-Procedure: Before the procedure, children will be informed about the study through the 'Child Consent Form,' and parents will be informed via the 'Informed Consent Form.' Both verbal and written consents will be obtained. Data for children and parents who agree to participate will be recorded by the researcher in the 'Child Patient Introductory Information Form.' The FPS-R (Faces Pain Scale-Revised) will be explained to the child, and they will be asked if they have any pain before the procedure. The child will be asked to mark their pain on the scale. The VAS (Visual Analog Scale) will be explained to the parents, and both the parent and the observer will evaluate the child's pain level before the procedure using the Visual Analog Scale. The Child Fear Scale will also be explained to both the child and the parent. The child will mark the level of fear they are feeling at that moment related to the blood collection procedure on the Child Fear scale. The parent and the observer will also rate the child's observed fear level. Afterward, a pulse oximeter will be placed on the child's finger, and their SpO2 and pulse will be recorded starting 1 minute before the procedure.

Guided Imagery Group: Children in the Guided Imagery group will be instructed to listen to an audio recording titled 'A Walk in the Forest' before the blood collection. It will be explained that the injection will take place while they are listening to the recording. The child will also be instructed to close their eyes, imagine the content of the recording, and focus on the sound, thus helping to distract their attention from the procedure. One minute before the blood collection, the child will wear headphones, and the audio recording will start.

Virtual Reality Glasses Group: In the Virtual Reality group, unlike the Guided Imagery group, the child will wear virtual reality glasses and watch a 'Walk in the Forest' video created with artificial intelligence.

Control Group: Children in the control group will only receive a routine blood collection procedure, and they will only be given an explanation related to the blood collection procedure.

Blood Collection Procedure: The blood collection for all children included in the study will be performed by an experienced clinical nurse. Immediately after the procedure begins, the pulse and oxygen saturation levels of children in all groups will be recorded in the 'Application Record Form.'

Post-Procedure: Immediately after the blood collection procedure (when the syringe is removed) and 1 minute later, pulse and oxygen saturation levels will be recorded in the 'Application Record Form.'

In the virtual reality glasses group, after the measurements, the virtual reality glasses will be removed from the children, and in the Guided Imagery group, the headphones will be removed from the children.

Immediately after the procedure, both the experimental and control group children will be asked to mark their pain and fear levels using the Faces Pain Scale-Revised and Child Fear Scales.

Parents and observers will assess the child's pain level and fear level during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 8 and 14 years old.
* Both the child and the parent must volunteer to participate in the study.
* The child and the parent must speak Turkish at a native level.
* The child must not have taken any medication with analgesic, antipyretic, or anti-inflammatory effects within the last 6 hours

Exclusion Criteria:

* The child has visual, hearing, or speech impairments.
* The child is illiterate.
* The child has a clinical condition that prevents the use of VR glasses or headphones.
* The child has an allergy to strawberries (mentioned in the guided imagery script) or a fear of forests or squirrels.
* The child has a disease that may cause chronic pain.
* The child has any auditory, mental, or neurological disability that could affect participation in the study

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Pain | 5 minutes before the procedure, 1 minute before the procedure, 1 minute after the procedure, 5 minutes after the procedure
  The Faces Pain Scale-Revised (FPS-R) is a self-report tool designed to assess acute pain intensity in children aged 4 to 16. It features six facial expressions ranging from neutral (score 0) to severe pain (score 10). Scores of 1-3 indicate mild pain, 4-6 moderate pain, and 7-10 severe pain. The scale is valid, reliable, widely used, and freely available for research or clinical use without special permission. In this study, FPS-R will be used to evaluate children's pain levels before and after injections in both experimental and control groups.
  The Visual Analogue Scale (VAS), developed in 1921 by Hayes and Patterson, is a 10 cm horizontal line marked from "no pain" to "unbearable pain." Participants mark their pain level on the line, and the pain score is calculated by measuring the distance from the "no pain" end. VAS will be used in this study to measure pre- and post-injection pain levels, as assessed by both parents and the researcher.
Fear | 5 minutes before the procedure, 1 minute before the procedure, 1 minute after the procedure, 5 minutes after the procedure
  Children's Fear Scale (CFS)
  The Children's Fear Scale (CFS) is used to measure children's fear and anxiety. In this method, a picture displaying five facial expressions rated from 0 to 4 is shown to the child. A score of 0 indicates no fear or anxiety, while a score of 4 indicates the highest level of fear and anxiety. This scale can be administered by both the researcher and the family to assess fear and anxiety before and during a procedure. In this study, the CFS will be used to evaluate the levels of fear in children from both the experimental and control groups before and after the blood collection procedure.

SECONDARY OUTCOMES:
Heart Rate | 5 minutes before the procedure, one minute before the procedure, During procedure, one minute after the procedure, five minutes after the procedure
  A finger-type pulse oximeter will be used to measure the children's heart rate values before, during, and after the blood collection procedure. These pulse oximeter devices can measure a child's oxygen saturation and pulse values without the need for invasive procedures.
Oxygen Saturation | 5 minutes before the procedure, one minute before the procedure, During procedure, one minute after the procedure, five minutes after the procedure
  A finger-type pulse oximeter will be used to measure the children's oxygen saturation values before, during, and after the blood collection procedure. These pulse oximeter devices can measure a child's oxygen saturation and pulse values without the need for invasive procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No